CLINICAL TRIAL: NCT01322308
Title: Effect of Pioglitazone on Endothelial Function in Premenopausal Women With Uncomplicated Systemic Lupus Erythematosus, a Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Effect of Pioglitazone on Endothelial Function in Premenopausal Women With Uncomplicated Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Heart Institute, Mexico (Other Government)
Collaborators: National Council of Science and Technology, Mexico (Other); Universidad Nacional Autonoma de Mexico (Other)
Responsible Party: Principal Investigator, Nacu Caracas Portilla, Juan Gabriel Juarez Rojas PhD, National Heart Institute, Mexico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 05-487
Record Dates: First submitted 2011-03-23; First posted 2011-03-24 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Systemic Lupus Erythematosus
Keywords: lupus; HDL particles; endothelial function; pioglitazone
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- sugar pill (Placebo Comparator): tablet similar to comparator
  Interventions: Drug: placebo
- pioglitazone (Active Comparator): 30 mg tablets QD (taken once daily)
  Interventions: Drug: pioglitazone

INTERVENTIONS:
Drug: pioglitazone — 30 mg tablet QD (taken once daily)
  Other Names: actos; zactos
  Arms: pioglitazone
Drug: placebo — tablet taken once a day
  Arms: sugar pill

SUMMARY:
The present study aims to investigate the effect of pioglitazone (30 mg/day) on endothelial function in premenopausal women with SLE (systemic lupus erythematosus). Patients with hypertension, endocrine, hepatic or renal diseases will not be included, or pregnant /breast feeding women. This is a randomized, double blind, placebo controlled study.

DETAILED DESCRIPTION:
SLE (systemic lupus erythematosus) is characterized by accelerated atherosclerosis. The risk of suffering an acute myocardial infarction among premenopausal women with SLE is 50 times higher than control women of the same age. Insulin resistance and hyperinsulinemia are frequent in SLE. Lipid metabolism in SLE, as in other insulin resistant states, is characterized by high triglycerides, low HDL-cholesterol, normal LDL cholesterol (or slightly increased) and an increase in LDL's susceptibility to oxidation.

All these alterations can produce endothelial dysfunction which is present in SLE patients. Pioglitazone is a PPAR (peroxisome proliferator activated receptor) gamma agonist that can potentially improve insulin resistance, with a positive effect on the lipid profile (lowering of triglycerides, and a discrete increase in HDL-C) and improve endothelial function.

Patients will be randomized to receive either placebo or pioglitazone 30 mg/day during a period of 12 weeks. Endothelial function will be assessed by Positron Emission Tomography (PET).

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants were premenopausal women with SLE
* Older than 18 years
* Attending the outpatient Rheumatology Clinic at three Mexico City community tertiary care hospitals

Exclusion Criteria:

* menopause
* diabetes
* thyroid dysfunction
* neurological
* hepatic
* renal or liver disease
* personal history of high blood pressure
* CHD (coronary heart disease)
* cerebrovascular events
* chronic or acute infections
* malignancy
* nor history of chronic drugs or alcohol abuse
* smoking
* pregnancy or breast-feeding
* intake of hormones or lipid-regulating drugs

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2007-03; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
improvement of endothelial function | 12 weeks
  Basal and final (12 weeks) endothelial function parameters measured by PET scan

SECONDARY OUTCOMES:
change in HDL particle physicochemical characteristics | 12 weeks
  HDL particle size, distribution and composition evaluated at baseline and at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Posadas, MD, Study Chair — Head of the Endocrinology Department

REFERENCES:
- [Derived] Juarez-Rojas JG, Medina-Urrutia AX, Jorge-Galarza E, Caracas-Portilla NA, Posadas-Sanchez R, Cardoso-Saldana GC, Goycochea-Robles MV, Silveira LH, Lino-Perez L, Mas-Oliva J, Perez-Mendez O, Posadas-Romero C. Pioglitazone improves the cardiovascular profile in patients with uncomplicated systemic lupus erythematosus: a double-blind randomized clinical trial. Lupus. 2012 Jan;21(1):27-35. doi: 10.1177/0961203311422096. Epub 2011 Oct 12. PMID 21993383